CLINICAL TRIAL: NCT05649462
Title: Retrospective Analysis of the Effect of Vitamin D Supplementation on the Clinical Efficacy of Vedelizumab in Ulcerative Colitis Patients
Brief Title: Effect of Vitamin D Supplementation on Vedolizumab Response in Patients With Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2022-07-27
Record Dates: First submitted 2022-10-24; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-10

CONDITIONS: Ulcerative Colitis; Vitamin D Deficiency; Vitamin D Supplement
MeSH Terms: conditions — Colitis, Ulcerative; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- supplementary group: take vitamin D supplementation (400 IU/day) during VDZ treatment
- non-supplementary group

SUMMARY:
It is uncertain whether vitD3 supplementation is beneficial for the remission of ulcerative colitis (UC). The effects of vitD3 supplements on the efficacy of vidrecizumab in Chinese UC patients were retrospectively analyzed. Methods: Patients with moderate to severe UC were recorded. These patients were initially treated with VDZ. VitD3 supplementation was defined as 400IU/d vitD3 supplementation during the first infusion of VDZ and continued throughout the follow-up period. Disease activity was assessed using the modified Mayo score.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe UC
* Treated with Vedolizumab

Exclusion Criteria:

* had recent supplementation of vitD3
* pregnant
* had cognitive/developmental disorders that affected their ability to complete the study procedures
* had medical illness or therapies potentially affecting bone, nutrition or growth status
* unknown or untested baseline serum 25(OH)D level

Ages: 15 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Serum 25 (OH) D level | 30 weeks
  Because serum 25 (OH) D levels are relatively stable, they are considered the most reliable indicator of vitamin D status.
disease activity | 30 weeks
  modified Mayo score，mild: 3 to 5, moderate: 6 to 10, severe: 11 to 12

SECONDARY OUTCOMES:
drug survival | 54 week
  Proportion of UC patients who continued to receive VDZ

CONTACTS AND LOCATIONS:
Overall Officials: Xia shenglong, Master, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China